CLINICAL TRIAL: NCT03793374
Title: The Efficacy of Modified Suction-assisted Cartilage Shaver for Axillary Osmidrosis
Brief Title: Modified Suction-assisted Cartilage Shaver for Axillary Osmidrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shang-Hung Lin, Attending physician of the Department of Dermatology of Kaohsiung Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Other Study IDs: 201801926B0
Record Dates: First submitted 2018-12-28; First posted 2019-01-04 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Treatment Outcome; Axillary Odor, Variation in
Keywords: Axillary osmidrosis; Surgery; Cartilage shaver

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Axillary osmidrosis patients: Patients with axillary malodor and require surgical intervention. The subcutaneous apocrine glands shaving were used.
  Interventions: Other: Subcutaneous apocrine glands shaving

INTERVENTIONS:
Other: Subcutaneous apocrine glands shaving — A 0.5-cm long incision was made in the identified elliptical surgical area at each axilla for the access of arthroscopy to remove the apocrine glands. A suction-assisted cartilage shaver (E9005 System, Linvatec Corporation, Largo, Florida, USA) was introduced through the incisions to remove of the subcutaneous apocrine glands radially. After defatting, the incisions were closed primarily with 4-0 polyglactin. We anchored the defatting skin to the axillary fascia by 4-0 nylon sutures instead of the tie-over dressing or tissue glues, and we also made several drainage holes by inserting an 18G needle obliquely into the defatting skin. Therefore, draining tubes were no longer needed. We will remove the stiches at the 8th day after the operation.

SUMMARY:
This study included patients who suffered from moderate to severe axillary osmidrosis to receive the modified suction-assisted cartilage shaver, and evaluated the efficacy and complications.

DETAILED DESCRIPTION:
<Patients> After obtaining the agreement of Chang Gung Medical Foundation Institutional Review Board, the investigators retrospectively included patients from July 2013 to September 2017. There were 39 patients treated for AO by the same dermatologist with suction-assisted cartilage shaver at the Department of Dermatology, Chang Gung Memorial Hospital, Kaohsiung, Taiwan. There were 28 females and 11 males, ranging from 14 to 52 years of age. The participants were all bothered by the axillary osmidrosis, which had a huge impact on their daily life with the embarrassing malodors. Operations were performed under local anaesthesia and in an outpatient basis.

<Operation> During the procedure, both of patient's axillae were exposed with the patient lying supine and arms abducted to avoid injury to the brachial plexus. The investigator cut the axillary hair short for better visualizing the region of apocrine glands, which are located near the hair follicles. The hair bearing elliptical region of axilla was marked before hair cutting. Tumescent solution was prepared with 0.1% lidocaine, 1:500,000 epinephrine and 10mEq/L sodium bicarbonate. The investigator injected the tumescent solution to the subcutaneous level of each axilla in view of the hydro-dissection ability of tumescent and minimizing the bleeding.

A 0.5-cm long incision was made in the center of identified elliptical surgical area at each axilla for the better access of arthroscopy to remove the apocrine glands located at dermo-subcutaneous junction, and for hiding the scar in the skin crease to make it less noticeable. A suction-assisted cartilage shaver (E9005 System, Linvatec Corporation, Largo, Florida, USA) was introduced through the incisions to remove of the subcutaneous tissue containing the apocrine glands radially. The investigator set the system to keep the inner cannula at 1500 rotations per minute in oscillation mode. After defatting, the incisions were closed primarily with 4-0 polyglactin. The investigator anchored the defatting skin to the axillary fascia by using 4-0 nylon sutures instead of the tie-over dressing used in the conventional shaver procedure, and the investigator also made several drainage holes by inserting an 18G needle obliquely into the defatting skin rather than placing the drainage tubes used in the conventional shaver procedure. Therefore, draining tubes were no longer needed. The investigator will remove the stitches at the 8th day after the operation.

<Efficacy assessments> The participants' medical history, physical examinations, and vital signs were carefully collected before the operation. The investigators retrospectively evaluated the pre- and post-operative clinical efficacies with a patient-centered scoring method. The severity of AO before the operation was classified from 1 to 5 to indicate the least severe to the most severe condition, from undetectable, mild, moderate, severe, to unbearable of malodor. The clinical efficacy was classified to 5 grades: poor (0%-20%), fair (21%-39%), acceptable (40%- 59%), good(60%-79%), and excellent (80%-100%), which was evaluated based on the elimination of malodor and the post-operative satisfaction. To evaluate the safety, adverse reactions such as hematoma, seroma, infection, wound necrosis, skin necrosis or perforation, and scar formation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe axillary osmidrosis and require surgical intervention.

Exclusion Criteria:

* Patients with bleeding tendency were excluded.
* Patients with active infections.
* Patients with major cardiovascular diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with axillary osmidrosis and require surgical intervention.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The change of malodor of axillary osmidorsis after the modified suction-assiated cartilage shaver | The treatment efficacy is evaluated 1 year after the surgery.
  The efficacy of surgical treatment for axillary osmidrosis is evaluated by the change of the malodor. The degree of malodor is subjective, therefore, the investigators classified the degree of malodor from 1 to 5 to indicate the least severe to the most sever condition. The degree of malodor was recorded before the operation, 1 month after the operation, and 1 year after the operation. The investigators evaluate the efficacy of the surgical treatment by the changes of the degree of the malodor of axillary osmidrosis.

SECONDARY OUTCOMES:
The rate of complications of the modified suction-assiated cartilage shaver for axillary osmidrosis | The immediate and longterm complications are recorded and evaluated at 1 week and 1 year respectively after the surgery.
  To evaluate the safety of the modified surgical method, adverse reactions such as hematoma, seroma, infection, wound necrosis, skin necrosis or perforation, and scar formation were recorded and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Hung Lin, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshikata R, Yanai A, Takei T, Shionome H. Surgical treatment of axillary osmidrosis. Br J Plast Surg. 1990 Jul;43(4):483-5. doi: 10.1016/0007-1226(90)90019-v. No abstract available. PMID 2393776
- [Background] Wu WH. Ablation of apocrine glands with the use of a suction-assisted cartilage shaver for treatment of axillary osmidrosis: an analysis of 156 cases. Ann Plast Surg. 2009 Mar;62(3):278-83. doi: 10.1097/SAP.0b013e3181776398. PMID 19240525
- [Background] Chern E, Yau D, Chuang FC, Wu WM. Arthroscopic shaver with refinement for axillary osmidrosis. Int J Dermatol. 2010 Jul;49(7):813-7. doi: 10.1111/j.1365-4632.2010.04540.x. PMID 20618505
- [Background] Lee JC, Kuo HW, Chen CH, Juan WH, Hong HS, Yang CH. Treatment for axillary osmidrosis with suction-assisted cartilage shaver. Br J Plast Surg. 2005 Mar;58(2):223-7. doi: 10.1016/j.bjps.2004.07.002. PMID 15710118
- [Derived] Tseng YJ, Lee CH, Lin SH. Modified Suction-Assisted Cartilage Shaver for Axillary Osmidrosis. Biomed Res Int. 2019 May 8;2019:7314753. doi: 10.1155/2019/7314753. eCollection 2019. PMID 31205944